CLINICAL TRIAL: NCT06488820
Title: Safety and Efficacy of Pulsed-field Ablation for Atrial Fibrillation in High Versus Low-volume Ablation Centers
Brief Title: Safety and Efficacy of Pulsed-field Ablation for Atrial Fibrillation in High Versus Low-volume Ablation Centers (SAFFICIENT)
Acronym: SAFFICIENT
Status: Terminated | Type: Observational
Why Stopped: Given the recent FDA approval of the VARIPULSE platform in November 2024, J&J MedTech and the PI have made the strategic decision to phase out SAFFICIENT IDE to focus on the post-approval study
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCAI_SAFFICIENT
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: pulsed-field ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Catheter ablation using pulsed-field ablation (PFA) system — PFA will be used to isolate the pulmonary veins and additional left atrial structure as needed

SUMMARY:
Catheter ablation using radiofrequency (RF) energy has been widely adopted for management of atrial fibrillation (AF) for the past several years.

However, heterogeneity of outcomes and complication rates are still reported that have been partly attributed to operator's experience and center's procedure volume (1). In a meta-analysis of 14 studies, both hospital volume of ≥50 and ≥100 procedures per year were associated with significantly lower complication rate compared to <50/year (2).

Pulse-field ablation (PFA) is an emerging technology for AF management that has demonstrated tremendous potential in terms of preferential tissue ablation with no damage to the adjacent organs. In the MANIFEST-PF survey, 24 European centers participated that had a mean of 704 ablations per year with 73.3 (range 7-291) PFA ablations annually (3). No post-PFA esophageal complications, PV stenosis or persistent phrenic nerve injury were reported. There appeared to be a trend toward fewer complications with center experience, particularly for pericardial tamponade (3).

However, the impact of number of PFA performed on procedure-success and safety has not been evaluated in the US.

This multicenter prospective study is designed to compare the incidence of adverse event (AE) and long-term procedural success of pulse-field ablation for AF in low volume (<100/year) vs. high volume (≥100/year) centers.

DETAILED DESCRIPTION:
Prospective, non-randomized, multi-center study NUMBER OF STUDY CENTERS: Up to 80 TRIAL OBJECTIVE To evaluate safety of the VARIPULSE™ Catheter when used in conjunction with the TRUPULSE™ Generator for catheter ablation in low volume centers, compared to high-volume centers, for the treatment of subjects with symptomatic atrial fibrillation, excluding long-standing persistent AF.

HYPOTHESIS The low volume centers would be noninferior to high volume centers with respect to the proportion of patients experiencing at least one primary adverse event (PAE).

ABLATION PROCEDURE All left atrial ablations such as pulmonary vein isolation (PVI) and isolation of left atrial posterior wall will be performed using the PFA system. If the right atrial structures are needed to be ablated (i.e. cavotricuspid isthmus line, coronary sinus), a commercially approved radiofrequency (RF) catheter and compatible RF generator will be used.

MANDATORY: Minimum applications per vein is 12, Maximum applications per vein is 20 Ablation Outside the PV

Ablation outside the PVs will be performed only in the presence of spontaneous triggers or documentation that those locations are the sites for triggers responsible for re-initiation of the arrhythmia either spontaneously or after isoproterenol challenge. For ablation outside the pulmonary vein, the number of applications will be determined on a case- by-case basis based on the expected tissue thickness in the ablation area. At a minimum, at least 6 applications per area (3 applications at 2 catheter rotations) should be considered. Each lesion set attempted will be assessed for acute efficacy (bi-directional block, absence of detectable electrograms). Additional lesions should be given until the acute endpoint is met.

Posterior wall ablations: Concentric overlapping ablations should be placed onto the posterior wall deliberately. The catheter will be rotated once between a pair of applications; briefly, rotation is performed such that, post-rotation, the splines are situated midway between the splines' pre- rotation positions. The number of applications will be at the operator's discretion.

DURATION OF SUBJECT PARTICIPATION:

11 months after the index ablation procedure (2 months blanking + 9 months follow-up)

DURATION OF STUDY 2-3 years (1-2 year of enrollment+ 11 months of study duration)

STATISTICS

The sample size and power calculation were performed to establish noninferiority (NI) of low volume centers with respect to the primary safety endpoint. With a NI margin of 0.04, an estimated sample size of 1084 patients per group will provide 80% power at one-sided significance level of 2.5% to declare non-inferiority. Considering 5% oversampling for attrition, 1138 patients will be enrolled per group.

Interim analysis: None planned

ELIGIBILITY:
Inclusion Criteria:

* Age: >≥18 years

  * Symptomatic Paroxysmal or Persistent AF patients of ≤ 1 year
  * First ablation or redo procedure to treat AF
  * Willing to provide written informed consent
  * Able and willing to comply with all testing and requirements

Exclusion Criteria:

* Long-standing persistent AF Page 17 of 70

  * Any condition contraindicating chronic anticoagulation
  * Prosthetic mechanical valves
  * Recent MI (in <3 months)
  * Active systemic infection
  * Pregnant or lactating women
  * Current enrollment in an investigational study evaluating another device or drug.
  * Documented left atrial (LA) thrombus by imaging within 48 hours before procedure (computed tomography (CT), transesophageal echocardiogram (TEE), or intracardiac echocardiogram (ICE) at the beginning of the procedure).
  * Uncontrolled heart failure or New York Heart Association (NYHA) Class IV
  * Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
  * Life expectancy less than 12 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Safety of PFA | 1 year
  Adverse events

SECONDARY OUTCOMES:
Efficacy of PFA | 2-mo blanking period+ 11 months
  Arrhythmia-free on- or off-antiarrhythmic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, Principal Investigator — Texas Cardiac Arrhythmia Institute, St.
Locations (1):
- Texas Cardiac Arrhythmia, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided